CLINICAL TRIAL: NCT01658891
Title: A SINGLE CENTRE, RANDOMISED, DOUBLE-BLIND, DOUBLE-DUMMY, 2-WAY CROSS OVER STUDY TO COMPARE SAFETY ASSESSED BY KNEMOMETRY AND URINARY CORTISOL MEASUREMENTS OF CHF1535 50/6 NEXThaler® (FIXED COMBINATION OF BECLOMETHASONE DIPROPIONATE AND FORMOTEROL FUMARATE) AND THE FREE COMBINATION OF LICENSED BECLOMETHASONE DIPROPIONATE AND FORMOTEROL FUMARATE IN ASTHMATIC CHILDREN ALREADY TREATED WITH INHALED CORTICOSTEROIDS
Brief Title: Comparison of Combination of Beclomethasone Dipropionate and Formoterol Fumarate Versus Single Components Assessed by Knemometry and Urinary Cortisol Measurements in Asthmatic Children
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-1110-PR-0071
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Asthma in Children
MeSH Terms: interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF 1535 50/6 µg (Experimental)
  Interventions: Drug: combination of beclomethasone dipropionate 50µg + formoterol fumarate 6µg
- beclomethasone dipropionate 100µg + Formoterol fumarate 6µg (Active Comparator)
  Interventions: Drug: free combination of beclomethasone dipropionate 100µg + Formoterol fumarate 6µg

INTERVENTIONS:
Drug: combination of beclomethasone dipropionate 50µg + formoterol fumarate 6µg — beclomethasone dipropionate 50µg + formoterol fumarate 6µg, 2 inhalations b.i.d. for 2 weeks
  Arms: CHF 1535 50/6 µg
Drug: free combination of beclomethasone dipropionate 100µg + Formoterol fumarate 6µg — beclomethasone dipropionate 100µg, 1 inhalation b.i.d. for 2 weeks and formoterol fumarate 6µg, 2 inhalations b.i.d. for 2 weeks
  Arms: beclomethasone dipropionate 100µg + Formoterol fumarate 6µg

SUMMARY:
single center, double-blind, double-dummy, 2-way cross over study in asthmatic children already treated with inhaled corticosteroids

ELIGIBILITY:
Inclusion Criteria:

* Prepuberal male and female outpatients, ≥ 5 and < 12 years old in Tanner stadium I according to Investigator's assessment;
* Clinical diagnosis of mild asthma during at least two months prior to screening visit;
* Forced Expiratory Volume during the first second (FEV1) > 80% of predicted normal values at screening visit;

Exclusion Criteria:

* Endocrinological diseases including growth impairment or other chronic diseases;
* Any concomitant disease requiring additional treatment with topic or systemic glucocorticosteroids;

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-11 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Lower Leg Growth rate measured by Knemometry | after 2 weeks of treatment

SECONDARY OUTCOMES:
24-hour urinary free cortisol/creatinine levels | after 2 weeks of treatment
Changes in pre-dose morning and evening PEF (L/min) | after 2 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- BørneAstmaKlinikken, Copenhagen, Denmark